CLINICAL TRIAL: NCT00543725
Title: A Phase III, Randomized, Double-blind Trial of TMC278 25mg q.d. Versus Efavirenz 600mg q.d. in Combination With a Background Regimen Containing 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors in Antiretroviral-naive HIV-1 Infected Subjects.
Brief Title: TMC278-TiDP6-C215: A Clinical Trial in Treatment Naive HIV-subjects Patients Comparing TMC278 to Efavirenz in Combination With 2 Nucleoside/Nucleotide Reverse Transcriptase Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR002704; TMC278-TIDP6-C215 (Other: Tibotec Pharmaceuticals, Ireland); NCT00614692 (obsolete NCT alias)
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Results first posted 2011-07-12 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections; HIV-1
Keywords: Antiretroviral; HIV-1; AIDS; TMC278-C215; TMC278-TiDP6-C215; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Rilpivirine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 002 (Active Comparator): efavirenz 600 mg tablet once daily for 96 weeks
  Interventions: Drug: efavirenz
- 001 (Experimental): TMC278 25 mg tablet once daily for 96 weeks
  Interventions: Drug: TMC278

INTERVENTIONS:
Drug: TMC278 — 25 mg tablet once daily for 96 weeks
  Arms: 001
Drug: efavirenz — 600 mg tablet once daily for 96 weeks
  Arms: 002

SUMMARY:
The purpose of this trial is to compare the effectiveness, safety and tolerability of TMC278 given at a dose of 25 mg once daily versus efavirenz (EFV) at a dose of 600 mg once daily, when combined with a background regimen containing 2 nucleoside/nucleotide reverse transcriptase inhibitors ( investigator choice of ABC/3TC, TDF/FTC or AZT/3TC) in HIV-1 infected patients who have not yet taken any anti-HIV drugs. The following evaluations will be done: antiviral activity, immunologic changes, and viral geno-/phenotype evolution, relationship of Pharmacokinetics (PK) and PK/Pharmacodynamics and Medical resource utilization and treatment adherence.

DETAILED DESCRIPTION:
Over the past decade, anti-human immunodeficiency virus (HIV) drugs have been introduced sequentially for use in the clinic. Currently, patients are routinely being treated with 3 or 4 drug combinations including nucleoside/tide analogue reverse transcriptase inhibitors (NRTIs/NtRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors (PIs), and/or fusion inhibitors. New potent antiretroviral (ARV) compounds that work in people whose HIV-1 virus is resistant to available drugs are urgently needed. This is a Phase III, randomized (study medication is assigned by chance), double-blind (neither the study physician nor the patient knows the name of the study assigned medication), double-dummy, active-controlled trial to compare the effectiveness, safety, and ability to tolerate TMC278 versus efavirenz (EFV). The study will last for 104 weeks which includes a screening period of 4 weeks, a 96-week treatment period, followed by a 4 week follow-up period. Patients will be randomly assigned (like tossing a coin) to TMC278 or to efavirenz in combination with two other anti-HIV drugs of the class nucleoside/nucleotide reverse transcriptase inhibitors. The hypothesis to be provided in this study is that the investigational drug TMC278 will perform just like efavirenz (EFV) in terms of antiviral effectiveness (i.e., suppressing of the plasma viral load to a level < 50 HIV-1 RNA (ribonucleic acid) copies/mL, in ARV-naïve HIV-infected patients. During the trial, patients' health will be monitored by physical examination, interview to assess health and well being, and laboratory testing on blood and urine samples. Experimental Group: One tablet of TMC278 25 mg daily; plus efavirenz (EFV) placebo; plus 2 nucleoside/nucleotide reverse transcriptase inhibitors; Control Group: One tablet of Placebo daily that looks just like TMC278 plus EFV 600 mg daily plus 2 nucleoside/nucleotide reverse transcriptase inhibitors for 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented HIV-1 infection
* Patient has never been treated with a therapeutic HIV vaccine or an ARV drug prior to screening
* Patient's HIV-1 plasma viral load at screening is > 5,000 HIV-1 RNA copies/mL (assayed by RNA PCR standard specimen procedure)
* Patient's virus is sensitive to the 2 nucleoside/nucleotide reverse transcriptase inhibitors chosen for treatment
* Patient agrees not to start ART before the baseline visit
* Patient is HLA-B*5701 negative in case abacavir is included in the patient's treatment regimen.

Exclusion Criteria:

* Previous use of ANY ARV drug for ANY length of time
* Any documented evidence of NNRTI resistance associated mutations in patient's HIV
* Category C AIDS defining illness, except, Stable Kaposi Sarcoma Wasting syndrome if not progressive
* Pneumocystis carinii pneumonia (PCP) that is considered not cured
* Active TB
* Allergy or hypersensitivity to study or background ARTs
* Specific grade 3 or 4 toxicity
* Kidney impairment: calculated creatinine clearance <50 ml/min

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (82):
- United States (25):
  - Long Beach, California
  - Los Angeles, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Newark, New Jersey
  - Flushing, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
- Australia (3):
  - Darlinghurst
  - Prahran
  - Surry Hills
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven
- Brazil (5):
  - Campinas
  - Distrito Barao Geraldo-Campina
  - Pinheiros
  - Recife
  - São Paulo
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto, Ontario
  - Montreal, Quebec
- Chile (2):
  - Providencia
  - Santiago
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai
- San José, Costa Rica
- France (4):
  - Clamart
  - Le Kremlin-Bicêtre
  - Montpellier
  - Paris
- Germany (7):
  - Berlin
  - Cologne
  - Essen
  - Frankfurt
  - Hamburg
  - Hanover
  - Mannheim
- India (2):
  - Chennai
  - Nagpur
- Mexico (2):
  - Guadalajara
  - Mexico City
- Panama City, Panama
- Porto, Portugal
- San Juan, Puerto Rico
- Russia (4):
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Voronezh
- South Africa (6):
  - Bloemfontein
  - Cape Town
  - Dundee
  - Johannesburg
  - Pretoria
  - Westdene Johannesburg Gauteng
- Spain (3):
  - Barcelona
  - Elche
  - Madrid
- Bangkok, Thailand
- United Kingdom (2):
  - London
  - Manchester

REFERENCES:
- [Derived] Rimsky L, Van Eygen V, Hoogstoel A, Stevens M, Boven K, Picchio G, Vingerhoets J. 96-Week resistance analyses of rilpivirine in treatment-naive, HIV-1-infected adults from the ECHO and THRIVE Phase III trials. Antivir Ther. 2013;18(8):967-77. doi: 10.3851/IMP2636. Epub 2013 May 28. PMID 23714781
- [Derived] Nelson M, Amaya G, Clumeck N, Arns da Cunha C, Jayaweera D, Junod P, Li T, Tebas P, Stevens M, Buelens A, Vanveggel S, Boven K; ECHO and THRIVE Study Groups. Efficacy and safety of rilpivirine in treatment-naive, HIV-1-infected patients with hepatitis B virus/hepatitis C virus coinfection enrolled in the Phase III randomized, double-blind ECHO and THRIVE trials. J Antimicrob Chemother. 2012 Aug;67(8):2020-8. doi: 10.1093/jac/dks130. Epub 2012 Apr 24. PMID 22532465
- [Derived] Cohen CJ, Andrade-Villanueva J, Clotet B, Fourie J, Johnson MA, Ruxrungtham K, Wu H, Zorrilla C, Crauwels H, Rimsky LT, Vanveggel S, Boven K; THRIVE study group. Rilpivirine versus efavirenz with two background nucleoside or nucleotide reverse transcriptase inhibitors in treatment-naive adults infected with HIV-1 (THRIVE): a phase 3, randomised, non-inferiority trial. Lancet. 2011 Jul 16;378(9787):229-37. doi: 10.1016/S0140-6736(11)60983-5. PMID 21763935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase III, randomized, double-blind trial of TMC278 25 mg q.d. versus efavirenz 600mg q.d. in combination with a background regimen containing 2 nucleoside/nucleotide reverse transcriptase inhibitors in antiretroviral-naïve HIV-1 infected subjects
Pre-assignment Details: 680 participants were randomized (340 in TMC 278 and 340 in efavirenz) but only 338 participants were treated with efavirenz (2 were randomized but not treated).
Groups:
- TMC278: 25 mg tablet once daily
- Efavirenz: 600 mg once daily
Period: Overall Study
Arm/Group | TMC278 | Efavirenz
Started | 340 | 338
Completed | 272 | 264
Not Completed | 68 | 74
Not completed — Adverse Event | 18 | 27
Not completed — Sponsor's Decision | 0 | 1
Not completed — Subject Non-Compliant | 4 | 4
Not completed — Subject Ineligible To Continue The Trial | 2 | 0
Not completed — Subject Reached A Virologic Endpoint | 22 | 14
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 13
Not completed — Lost to Follow-up | 15 | 11
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC278 | Efavirenz | Total
Number analyzed (Participants) | 340 | 338 | 678
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 339 | 337 | 676
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (9.39) | 36.4 (8.92) | 36.5 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 94 | 184
  Male | 250 | 244 | 494
Region Enroll [Number; unit: participants]
  Africa | 19 | 38 | 57
  Asia | 59 | 61 | 120
  Latin America | 90 | 85 | 175
  USA, Canada, Europe, Australia | 172 | 154 | 326

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <50 Copies Per mL) at Week 48
Description: Virological response is defined as confirmed plasma viral load less than (<) 50 human immunodeficiency virus-1 (HIV-1) (ribonucleic acid [RNA]) copies/milliliter (ml) at Week 48. The TLOVR algorithm was used to derive response. Response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders after discontinuation. Resuppression after confirmed virologic failure was considered as failure. Virologic Failure includes participants who were rebounder (confirmed viral load >= 50 copies/ml after being responder) or who were never suppressed (no confirmed viral load <50 copies/ml).
Time Frame: Week 48
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 340 | 338
Participants
  Responder | 291 | 276
  Virologic failure | 24 | 18
  Death | 1 | 3
  Discontinued due to AE | 8 | 21
  Discontinued due to other reason than AE | 16 | 20
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Assuming a response rate of 75% at 48 weeks for both treatment groups, 340 subjects were needed per treatment (TMC278 or EFV) to establish non-inferiority of TMC278 versus EFV with a maximum allowable difference of 12% and a 1-sided significance level of 2.5%, to yield 95% power; Test type: Non-Inferiority or Equivalence — If the lower limit of the 95% 2-sided confidence interval of the difference in proportions (TMC278 - EFV) exceeds -12%, non-inferiority of TMC278 versus EFV can be concluded; p < 0.0001, Regression, Logistic — Significance level was set at 2.5% (one-sided). No adjustment of p-value for multiple comparisons, since there was only single comparison for the primary endpoint; Logistic regression model included treatment arm and background NRTI regimen as factors, and baseline (log10) viral load as covariate; Difference in proportion of response = 3.7, 95% CI [-1.6 to 9.0] — Difference in proportion responders was estimated through the logistic regression model

2. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Snapshot, <50 Copies Per mL) at Week 48
Description: The analysis is based on the last observed viral load (VL) data within the Week 48 window. Virologic response is defined as a VL<50 copies/mL (observed case). Missing VL was considered as non-response. Virologic Failure includes subjects who had VL>=50 copies/mL in the Wk 48 window, subjects who discontinued early due to lack or loss of efficacy, subjects who discontinued for reasons other than an adverse event, death or lack or loss of efficacy and at the time of discontinuation had a VL>=50 copies/mL and subjects who had a switch in background regimen that was not permitted by the protocol.
Time Frame: Week 48
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 340 | 338
Participants
  Virologic Response (<50 copies/mL) | 281 | 265
  Virologic failure | 41 | 38
  No plasma viral load data in 48-week window | 18 | 35
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Difference in proportion of response = 3.9, 95% CI [-1.9 to 9.6] — Difference in proportion responders was estimated through the logistic regression model

3. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <50 Copies Per mL) at Week 96
Time Frame: Week 96
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 340 | 338
Participants
  Responder | 269 | 258
  Virologic failure | 34 | 24
  Death | 1 | 3
  Discontinued due to AE | 16 | 23
  Discontinued due to other reason than AE | 20 | 30
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in proportion of response = 2.4, 95% CI [-3.6 to 8.4] — Difference in proportion responders was estimated through the logistic regression model

4. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Snapshot, <50 Copies Per mL) at Week 96
Time Frame: Week 96
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 340 | 338
Participants
  Virologic response (<50 copies/mL) | 259 | 254
  Virologic failure | 53 | 38
  No plasma viral load data in 96-Week window | 28 | 46
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Difference in proportion of response = 0.7, 95% CI [-5.6 to 7.0] — Difference in proportion responders was estimated through the logistic regression model

5. Secondary Outcome: Number of Participants With Virological Response (Observed, <50 Copies/mL) at Last On-Treatment Visit (Post-Week 96).
Description: Virological response is defined as (observed) plasma viral load less than 50 human immunodeficiency virus-type 1 (HIV-1) ribonucleic acid (RNA) copies per mL at the last on-treatment post-Week 96 visit.
Time Frame: Variable, ranging from 3 months up to maximum 18 months for TMC278 and 12 months for Efavirenz
Population: Participants with at least 1 Post-Week 96 visit were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 269 | 257
Participants | 260 | 246

6. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <400 Copies Per mL) at Week 48
Description: Virological response is defined as confirmed plasma viral load < 400 HIV-1 (RNA) copies/mL at Week 48. The TLOVR algorithm was used to derive response. Response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders after discontinuation. Resuppression after confirmed virologic failure was considered as failure. Virologic Failure includes participants who were rebounder (confirmed viral load >= 400 copies/mL after being responder) or who were never suppressed (no confirmed viral load <400 copies/mL).
Time Frame: Week 48
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 340 | 338
Participants | 300 | 286

7. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <400 Copies Per mL) at Week 96
Description: Virological response is defined as confirmed plasma viral load < 400 HIV-1 (RNA) copies/mL at Week 96. The TLOVR algorithm was used to derive response. Response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders after discontinuation. Resuppression after confirmed virologic failure was considered as failure. Virologic Failure includes participants who were rebounder (confirmed viral load >= 400 copies/mL after being responder) or who were never suppressed (no confirmed viral load <400 copies/mL).
Time Frame: Week 96
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 340 | 338
Participants | 283 | 270

8. Secondary Outcome: Mean Change From Baseline to Week 48 and Week 96 in Absolute and Relative CD4+ Cell Counts (Using Imputed Data)
Description: Change from baseline in CD4+ cell count was imputed in case of missing values: in case of premature discontinuation, data were imputed with the baseline value after discontinuation (i.e. change=0, Non-Completer [NC] = Failure); otherwise last observation carried forward was applied.
Time Frame: Baseline, Week 48, and Week 96
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Mean (95% Confidence Interval); unit: cells per microliter
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 339 | 338
cells per microliter
  Absolute cell count, Week 48 | 188.6 [173.98 to 203.15] | 170.7 [154.55 to 186.77]
  Absolute cell count, Week 96 | 234.5 [217.40 to 251.55] | 212.0 [193.70 to 230.34]
  Relative cell count, Week 48 | 8.3 [7.68 to 8.85] | 8.0 [7.39 to 8.60]
  Relative cell count, Week 96 | 10.1 [9.35 to 10.75] | 9.7 [8.95 to 10.40]

9. Secondary Outcome: Number of Participants With Virologic Failure for the Resistance Determinations by Developing Mutations: First Available On-Treatment Genotypic Data After Failure
Description: Virologic failure for the resistance determinations was defined as lack of virologic response (never having had 2 consecutive plasma viral load <50 copies/mL) and plasma viral load increase of >=0.5 log 10 copies/mL above nadir (i.e., never suppressed), or confirmed loss of virologic response (2 consecutive plasma viral load >=50 copies/mL after having had 2 consecutive plasma viral load <50 copies/mL; i.e., rebounder), or discontinued with a last observed on-treatment plasma viral load >=50 copies/mL after having had 2 consecutive plasma viral load <50 copies/mL. For this study, treatment-emergent reverse transcriptase (RT) resistance associated mutations (RAMs) occurring in at least 2 virologic failures (for at least one treatment group) for the following lists are presented: i) Extended list of Non-nucleoside reverse transcriptase inhibitor (NNRTI RAMs) ii) IAS-USA list of Nucleoside/tide reverse transcriptase inhibitor (N[t]RTI RAMs).
Time Frame: Week 96
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set. Here "N" (Number of Participants Analyzed) signifies number of Participants who were evaluable (had data) for this outcome.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 34 | 24
Participants
  Treatment-emergent NNRTI RAM | 17 | 11
  E138K | 13 | 1
  H221Y | 3 | 0
  K101E | 3 | 2
  K103N | 0 | 6
  V90I | 2 | 1
  V106M | 0 | 2
  V189I | 2 | 0
  Y188C | 0 | 2
  Treatment-emergent N(t)RTI RAM | 17 | 6
  K65R | 0 | 2
  K219E | 2 | 0
  M184I | 8 | 1
  M184V | 10 | 3

ADVERSE EVENTS:
Time Frame: Up to 164 weeks for participants in the TMC278 treatment group and up to 144 weeks for participants in the efavirenz treatment group.
Description: Only participants who had at least one of the treatment-emergent adverse events (TEAEs) listed in the Other (non Serious) adverse event (AE) table are included in the total number of participants with Non-Serious AEs.
Arm/Group | TMC278 | Efavirenz
Serious Adverse Events (participants affected / at risk) | 32/340 | 31/338
Other Adverse Events (participants affected / at risk) | 253/340 | 259/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC278 (N=340) | Efavirenz (N=338)
Pneumonia (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Cyclosporidium infection (Infections and infestations) | 0 | 1
Dysentery (Infections and infestations) | 0 | 1
Encephalitis herpes (Infections and infestations) | 0 | 1
Hepatitis c (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Jejunitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 2
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Food allergy (Immune system disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Brain scan abnormal (Investigations) | 1 | 0
Blood amylase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Macular hole (Eye disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Arthritis gonococcal (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
External ear cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Hepatitis b (Infections and infestations) | 1 | 0
Secondary syphilis (Infections and infestations) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC278 (N=340) | Efavirenz (N=338)
Nasopharyngitis (Infections and infestations) | 50 | 47
Upper respiratory tract infection (Infections and infestations) | 43 | 37
Bronchitis (Infections and infestations) | 31 | 6
Influenza (Infections and infestations) | 32 | 30
Pharyngitis (Infections and infestations) | 20 | 14
Headache (Nervous system disorders) | 61 | 53
Dizziness (Nervous system disorders) | 42 | 111
Somnolence (Nervous system disorders) | 17 | 28
Nausea (Gastrointestinal disorders) | 57 | 67
Diarrhoea (Gastrointestinal disorders) | 49 | 53
Vomiting (Gastrointestinal disorders) | 22 | 26
Insomnia (Psychiatric disorders) | 38 | 21
Abnormal dreams (Psychiatric disorders) | 19 | 26
Depression (Psychiatric disorders) | 24 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 15
Fatigue (General disorders) | 20 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 30
Rash (Skin and subcutaneous tissue disorders) | 15 | 49
Pyrexia (General disorders) | 15 | 17
Anogenital warts (Infections and infestations) | 17 | 14
Sinusitis (Infections and infestations) | 17 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 17
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 17
Hypertension (Vascular disorders) | 23 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days